CLINICAL TRIAL: NCT06312254
Title: Pharmacological Modulation of Peripheral Nerve Excitability - Measurement With the Human Perception Threshold Tracking Method
Brief Title: Pharmacological Modulation of Peripheral Nerve Excitability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Carsten Dahl Mørch, M.Sc., Ph.D., Associate Professor, Aalborg University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: N-20230071
Record Dates: First submitted 2024-02-27; First posted 2024-03-15 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Peripheral Neuropathy
Keywords: Topical treatment; Small fiber excitability; Perception Threshold Tracking Method
MeSH Terms: conditions — Peripheral Nervous System Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Participant and investigator/project involved personal is blinded to which cream is applied.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Pharmacological modulation with lidocaine 5% (Active Comparator): Experimental investigation of pharmacological modulation of peripheral nerve excitability, which is measured with the human perception threshold tracking method. With this method neurophysiological mechanisms of sensory afferents can be investigated
  Interventions: Drug: Topical lidocaine 5%
- Pharmacological modulation with Phenytoin 10% (Active Comparator): Experimental investigation of pharmacological modulation of peripheral nerve excitability, which is measured with the human perception threshold tracking method. With this method neurophysiological mechanisms of sensory afferents can be investigated
  Interventions: Drug: Topical Phenytoin 10%
- Pharmacological modulation with Mepyramine 2% (Active Comparator): Experimental investigation of pharmacological modulation of peripheral nerve excitability, which is measured with the human perception threshold tracking method. With this method neurophysiological mechanisms of sensory afferents can be investigated
  Interventions: Drug: Topical Mepyramine 2%
- Control (Placebo Comparator): Experimental investigation of pharmacological modulation of peripheral nerve excitability, which is measured with the human perception threshold tracking method. With this method neurophysiological mechanisms of sensory afferents can be investigated
  Interventions: Other: Topical Placebo

INTERVENTIONS:
Drug: Topical lidocaine 5% — Drug is used to pharmacologically modulate peripheral sensory afferents
  Arms: Pharmacological modulation with lidocaine 5%
Drug: Topical Phenytoin 10% — Drug is used to pharmacologically modulate peripheral sensory afferents
  Arms: Pharmacological modulation with Phenytoin 10%
Drug: Topical Mepyramine 2% — Drug is used to pharmacologically modulate peripheral sensory afferents
  Arms: Pharmacological modulation with Mepyramine 2%
Other: Topical Placebo — Drug is used as control
  Arms: Control

SUMMARY:
The present project is a human experimental study. The aim is to assess the pharmacologically modulated excitability of peripheral sensory nerves with a human experimental model.

The study measures the excitability of peripheral sensory nerves before and after application of different topical drugs (lidocaine (5%), phenytoin (10%),mepyramine (2%) and placebo).

DETAILED DESCRIPTION:
Design and method Study design The study is a randomized, double-blinded, placebo-controlled study. To minimize the risk of bias and achieve balance in the allocation of participants and application of creams, block randomization is used. To ensure double blinding, 1-2 colleagues from Center for Neuroplasticity and Pain (CNAP), who is not otherwise involved in the project, will keep the randomization list in a secure room.

Study procedure and experimental test The PTT model will be used to measure the excitability of peripheral sensory afferents. PTT will be measured before and after topical drug application at four distinct areas - two at each side of the volar site of the forearms.

In total four topical creams will be used in the study. One cream containing placebo, one with lidocaine (5%), one with phenytoin (10%) and one with mepyramine (2%).

The study consists of one session lasting 3-4 hrs. The study will include 20 healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Men and Women age > 18 years
* Understand and speak Danish
* No medication besides contraceptives

Exclusion Criteria:

* Pregnancy or lactating women
* Drug addiction (use of cannabis, opioids, or other drugs)
* Use of pain killers, alcohol, or nicotine within the last 24 hours before study start
* Any other medical treatment (e.g., antidepressants, anticonvulsants)
* History of peripheral or chronic pain conditions / neuropathy
* Skin diseases
* Scars and/or tattoos at the volar site of the forearm
* Previous traumatic experience of an electrical accident
* Application of moisturizing lotion of the volar site of the forearms (24 hours before study start)
* Participation in any other research projects/studies 7 days before study start
* Known allergy/intolerance to lidocaine/phenytoin/mepyramine
* Lack of ability to cooperate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-04-09 (Actual); Primary Completion 2024-12-02 (Actual); Study Completion 2024-12-11 (Actual)

PRIMARY OUTCOMES:
Change in PTT-value | 1 hour after application of cream
  Primary outcome measures are changes in the PTT-value (registered as mA) before and after application with topical pharmaceutical drugs.

CONTACTS AND LOCATIONS:
Overall Officials: Trine Andresen, Post.Doc, Study Director — Center for Neuroplasticity and Pain
Locations (1):
- Center for Neuroplasticity and Pain, Aalborg, Denmark